CLINICAL TRIAL: NCT02051166
Title: A Non Interventional, Retrospective Study on AECOPD Treatment Status in China
Brief Title: Clinical Practice of AECOPD Management in China
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-RCN-XXX-2013/1
Record Dates: First submitted 2014-01-24; First posted 2014-01-31 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-06

CONDITIONS: Acute Exacerbation of Chronic Obstructive Pulmonary Disease

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is observe clinical practice including glucocorticoids treatment in AECOPD in China.

DETAILED DESCRIPTION:
It is widely recognized that the global social and economic burden of Chronic obstructive pulmonary disease (COPD) is high; affecting an estimated 64 million people worldwide. It was reported the prevalence of COPD in China population over 40 years old is about 8.2% (Zhong Nanshan et al, 2007). According to the report on China Chronic Disease, COPD is the second disease of Disability Adjusted Life Years. The economic burden of COPD is tremendous in China. Cost analysis in 2006 showed that every COPD patient in urban would pay 1732.24 $ on medical cost every year, indirect cost on nurse and traffic is 231.6 $, total cost would account for 40% of average family income in 2006(Chiang CH.,2008).AECOPD is one of most important cause leading to COPD death. Corticosteroid is essential for AECOPD management and recommended by domestic and international guidelines. But it shows that corticosteroid use for treating AECOPD in China is around 70% from market research in big hospitals, and less report about how steroid is used for AECOPD management was published, including distribution, dosage, treatment duration, etc. The healthcare resources utilization for treating AECOPD in China is also unclear.

ELIGIBILITY:
Inclusion Criteria:

1. ≥40 years old
2. Hospitalization treatment due to AECOPD since Sep, 2013
3. Diagnosed by GOLD 2013 as COPD at least 3 months before AECOPD based on treating physician's judgment
4. Provided informed consent or informed consent waiver

Exclusion Criteria:

1. Participation in any interventional clinical study within 3 months before being recruited in the study.
2. Ongoing AECOPD during recruitment timeline
3. The patients whose symptoms haven't recovered and then discharge by themselves
4. The primary diagnosis of hospitalization is not AECOPD

Ages: 40 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient population will be ≥40 years of age, received hospitalization due to AECOPD since Sep, 2013. The patients should be diagnosed by GOLD 2013 as COPD at least 3 months before AECOPD based on treating physician judgment.
Sampling Method: Non-Probability Sample
Enrollment: 5095 (Actual)
Dates: Start 2014-02; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Percentage of glucocorticoids treatment for AECOPD | day 1 to up to 30 days (Hospital discharge)

SECONDARY OUTCOMES:
Percentage of oral /intravenous/ inhaled steroid therapy in patients treated with glucocorticoids, mean dosage, regimen and treatment duration via different administration route in hospital | day 1 to up to 30 days (Hospital discharge)
Percentage of antibiotics treatment for AECOPD by clinicians during the hospitalization. | day 1 to up to 30 days (Hospital discharge)
Mortality caused by AECOPD and recorded as primary cause of death by clinicians | day 1 to up to 30 days (Hospital discharge)
Percentage of antibiotics treatment via different administration route for AECOPD, mean treatment duration via different administration route in hospital | day 1 to up to 30 days (Hospital discharge)
Endotracheal intubation rate in treatment of AECOPD | day 1 to up to 30 days (Hospital discharge)
Pneumonia rate at the diagnose of AECOPD and in treatment of AECOPD | day 1 to up to 30 days (Hospital discharge)
Hospitalization duration and treatment cost due to AECOPD as primary cause | day 1 to up to 30 days (Hospital discharge)
Percentage of treatment category before AECOPD and at discharge | day 1 to up to 30 days (Hospital discharge)
Clinical efficacy and safety within different administration route of corticosteroid treatment | day 1 to up to 30 days (Hospital discharge)

OTHER OUTCOMES:
Demographic data | day 1
Year of COPD diagnosis | day 1
Any other significant medical condition or co-morbidities | day 1
Smoking status (number of pack-years) | day 1
Onset date of this AECOPD, date of hospitalization, date of discharge | day 1 to up to 30 days (Hospital discharge)

CONTACTS AND LOCATIONS:
Overall Officials: Wanzhen Yao, Ph.D, Principal Investigator — Peking University Third Hospital
Locations (13):
- China (13):
  - Research Site, Hefei, Anhui
  - Research Site, Beijing, Beijing Municipality
  - Research Site, Langfang, Hebei
  - Research Site, Baotou, Inner Mongolia
  - Research Site, Hohhot, Inner Mongolia
  - Research Site, Yinchuan, Ningxia
  - Research Site, Shanghai, Shanghai Municipality
  - Research Site, Taiyuan, Shanxi
  - Research Site, Xi’an, Shanxi
  - Research Site, Beijing
  - Research Site, Guangzhou
  - Research Site, Shanghai
  - Research Site, Tianjin

REFERENCES:
- [Derived] Zheng JP, Zhang J, Ma LJ, Chen P, Huang M, Ou XM, Zhao ZW, Jiang SJ, Cao J, Yao W. Clinical Outcomes Of Using Nebulized Budesonide As The Initial Treatment For Acute Exacerbations Of Chronic Obstructive Pulmonary Disease: A Post-Hoc Analysis. Int J Chron Obstruct Pulmon Dis. 2019 Nov 29;14:2725-2731. doi: 10.2147/COPD.S196615. eCollection 2019. PMID 31819404
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=2815&filename=NIS-RCN-XXX-2013_1_CSR_Synopsis.pdf
- See also: Yao et al AECOPD NIS abstract_2015 APSR abstract ID: 285 — http://onlinelibrary.wiley.com/doi/10.1111/resp.12706/epdf